CLINICAL TRIAL: NCT05990400
Title: Effectiveness and Safety of Topical Finasteride and Minoxidil Combination Compared to Topical Minoxidil for The Treatment of Male Androgenetic Alopecia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Farah Faulin Al Fauz Lubis, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23030293
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Androgenetic Alopecia
Keywords: Finasteride topical; Minoxidil topical; Male androgenetic alopecia
MeSH Terms: conditions — Alopecia | interventions — Finasteride; Minoxidil

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomized to receive either combination of minoxidil 5% topical and finasteride 0,1% topical or minoxidil 5% topical. The allocation sequence was generated with a computer by an analyst.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) The allocation sequence was generated with a computer by an analyst. The allocation sequence was concealed from the investigators, outcomes assessor, and subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of minoxidil 5% topical and finasteride 0,1% topical group (Experimental): Combination of minoxidil 5% solutio and finasteride 0,1% solutio which has administered topically
  Interventions: Drug: Finasteride; Drug: Minoxidil
- Minoxidil 5% topical group (Active Comparator): Minoxidil 5% solutio which has administered topically
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Finasteride — finasteride topical 0,1%
  Arms: Combination of minoxidil 5% topical and finasteride 0,1% topical group
Drug: Minoxidil — minoxidil topical 5%

SUMMARY:
A double-blind, randomized, controlled trial of 40 male patients with androgenetic alopecia was conducted. All subject were randomized to receive either combination of minoxidil 5% topical and finasteride 0,1% topical or minoxidil 5% topical

DETAILED DESCRIPTION:
All subject were randomized to receive either combination of minoxidil 5% topical and finasteride 0,1% topical or minoxidil 5% topical The primary outcome was increase of the hair density and hair diameter (mean thickness) measured by trichoscan Measurements were done at baseline and every four weeks for twelve weeks. Additionally, side effects of therapy was also measured.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged from 18-59 years diagnosed with androgenic alopecia
2. Androgenic alopecia type III-V according to Hamilton-Norwood criteria
3. Willing to participate in this research by signing the consent form after receiving an explanation from the researcher
4. Willing to not cutting the hair nor coloring the hair during the study

Exclusion Criteria:

1. Diagnosed with other infectious or inflammatory skin disease in the scalp
2. Using oral medications or vitamins that aim to increase the amount of hair in the last 1 month
3. Using topical medication that aim to increase the amount of hair in the last 2 weeks
4. Undergoing cosmetic procedure for AGA therapy such as low-level laser therapy (LLLT) procedures, platelet-rich plasma (PRP) injections, or microneedling within the last 3 months
5. Have sexual disorder such as decreased libido
6. Have a history of allergy or irritant contact dermatitis to the minoxidil and finasteride

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Hair density | 4 times of measurement in 3 months
  Density of the hair is the number of hair strands per square inch of the scalp measured by trichoscan
Hair diameter (mean thickness) | 4 times of measurement in 3 months
  Hair diameter is the midline of the hair shaft measured by trichoscan
Side effects | 4 times of measurement in 3 months
  Incidence of side effects

SECONDARY OUTCOMES:
Velus hair percentage ( hair rate vellus) | 4 times of measurement in 3 months
  Vellus hair is a hair that is less than 30 micrometer in diameter, lacks a medulla hair, and is 2 cm in length measured by trichoscan
Terminal hair percentage (hair rate terminal) | 4 times of measurement in 3 months
  Terminal hair is a hair that has a hair more than 60 micrometer, contains the medulla and can be up to 100 cm in length measured by trichoscan
Dermoscopy | 4 times of measurement in 3 months
  Dermoscopy is a non-invasive technique that allows more detailed examination of the scalp and hair shaft under magnification

CONTACTS AND LOCATIONS:
Locations (1):
- University Indonesia, Jakarta, Other (Non U.s.), Indonesia

IPD SHARING:
Plan to Share IPD: No